CLINICAL TRIAL: NCT04340362
Title: A Phase 2a, Open-label, Single-arm, 2-Part Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of VX-147 in Adults With APOL1-mediated Focal Segmental Glomerulosclerosis
Brief Title: Phase 2a Study of VX-147 in Adults With APOL1-mediated Focal Segmental Glomerulosclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX19-147-101; 2020-000185-42 (EudraCT Number)
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Results first posted 2023-07-10 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Glomerulosclerosis, Focal Segmental
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VX-147 (Experimental): All participants received VX-147 at a dosage of 15 mg once daily (qd) for 2 weeks and VX-147 at a dosage of 45 mg qd for 11 weeks. Part A was enrolled in 2 cohorts: Cohort 1 and Cohort 2. Cohort 1 included participants with urine protein to creatinine ratio (UPCR) approximately greater than or equal to (≥) 3 g/g (± 10%) and less than (<) 10 g/g and estimated glomerular filtration rate (eGFR) approximately ≥30 mL/min/1.73 m2 (± 10%). Cohort 2 included participants with UPCR approximately ≥0.8 g/g (± 10%) and <2.7 g/g and eGFR approximately ≥30 mL/min/1.73 m2.
  Interventions: Drug: VX-147

INTERVENTIONS:
Drug: VX-147 — Tablets for oral administration.
  Other Names: IXP

SUMMARY:
This study will evaluate the efficacy, safety and pharmacokinetics (PK) of VX-147 in participants with apolipoprotein L1 (APOL1)-mediated focal segmental glomerulosclerosis (FSGS).

ELIGIBILITY:
Key Inclusion Criteria:

* APOL1 genotype of G1/G1, G2/G2, or G1/G2
* FSGS diagnosed by kidney biopsy

Key Exclusion Criteria:

* Evidence of non-APOL1-mediated FSGS
* Participants with known sickle cell disease
* Solid organ or Bone marrow transplant

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-12-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (33):
  - University of Alabama at Birmingham - The Kirklin Clinic, Birmingham, Alabama
  - California Institute of Renal Research, San Diego, California
  - The George Washington University Medical Faculty Associates - Kidney Disease & Hypertension, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Kidney and Hypertension Specialists of Miami, Miami, Florida
  - Florida Premier Research Institute, Winter Park, Florida
  - Morehouse School of Medicine, Grady Memorial Hospital, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Georgia Nehphrology, Lawrenceville, Georgia
  - Central Georgia Kidney Specialists PC, Macon, Georgia
  - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Medical Center - New Orleans, New Orleans, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Renal and Transplant Associates of New England, PC, Springfield, Massachusetts
  - Paragon Health, PC d/b/a Nephrology Center, PC, Kalamazoo, Michigan
  - Nephrology and Hypertension Associates, LTD, Tupelo, Mississippi
  - St Louis Kidney Care, St Louis, Missouri
  - Nevada Kidney Disease and Hypertension Centers, Las Vegas, Nevada
  - SUNY Downstate, Brooklyn, New York
  - Urban Family Practice, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - UNC Kidney Center Division of Nephrology & Hypertension, Chapel Hill, North Carolina
  - Tryon Medical Partners, Charlotte, North Carolina
  - Durham Nephrology Associates, PA, Durham, North Carolina
  - Duke University School of Medicine - Duke Molecular Physiology Institute, Durham, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - South Carolina Nephrology and Hypertension Center, Inc., Orangeburg, South Carolina
  - Vanderbilt University VU, Nashville, Tennessee
  - Prolato Clinical Research Center, Houston, Texas
  - Privia Medical Group, Houston, Texas
- France (6):
  - Hopital Henri Mondor, Créteil
  - Hôpital Bicêtre AP-HP, Le Kremlin-Bicêtre
  - Bichat Hospital, Paris
  - Hopitaux Universitaires Est Parisien - Hopital Tenon, Paris
  - Service de Nephrologie - Hopital Universitaire Necker, Paris
  - Université Paris-Descartes / Hôpital Européen Georges Pompidou, Paris
- GCM Medical Group, PSC, San Juan, Puerto Rico
- United Kingdom (4):
  - University Hospitals of Leicester NHS Trust - Leicester General Hospital, Leicester
  - Barts Health NHS Trust, London
  - The Medicines Evaluation Unit, Manchester
  - King's College Hospital NHS Foundation Trust - Guthrie Clinic, Southwark

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent research/clinical-trial-data-sharing.

REFERENCES:
- [Derived] Egbuna O, Zimmerman B, Manos G, Fortier A, Chirieac MC, Dakin LA, Friedman DJ, Bramham K, Campbell K, Knebelmann B, Barisoni L, Falk RJ, Gipson DS, Lipkowitz MS, Ojo A, Bunnage ME, Pollak MR, Altshuler D, Chertow GM; VX19-147-101 Study Group. Inaxaplin for Proteinuric Kidney Disease in Persons with Two APOL1 Variants. N Engl J Med. 2023 Mar 16;388(11):969-979. doi: 10.1056/NEJMoa2202396. PMID 36920755
- [Derived] Bruggeman LA, Sedor JR, O'Toole JF. Apolipoprotein L1 and mechanisms of kidney disease susceptibility. Curr Opin Nephrol Hypertens. 2021 May 1;30(3):317-323. doi: 10.1097/MNH.0000000000000704. PMID 33767059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was planned in 2 parts: Part A (Treatment Period), which consisted of 2 cohorts (i.e., cohort 1 and 2) and Part B (Optional Exploratory Off-treatment Follow-up Period). The primary and secondary efficacy analyses and safety analyses were planned for only Part A.
Pre-assignment Details: This study was conducted on adult participants who had APOL1-mediated focal segmental glomerulosclerosis (FSGS).
Groups:
- VX-147: All participants received VX-147 at a dosage of 15 mg once daily (qd) for 2 weeks and VX-147 at a dosage of 45 mg qd for 11 weeks. Part A was enrolled in 2 cohorts: Cohort 1 and Cohort 2. Cohort 1 included participants with urine protein to creatinine ratio (UPCR) approximately greater than or equal to (≥) 3 g/g (± 10%) and <10 g/g and estimated glomerular filtration rate (eGFR) approximately ≥30 mL/min/1.73 m2 (± 10%). Cohort 2 included participants with UPCR approximately ≥0.8 g/g (± 10%) and <2.7 g/g and eGFR approximately ≥30 mL/min/1.73 m2.
Period: Overall Study
Arm/Group | VX-147
Started | 16
Cohort 1 (The milestone represents the number of participants in Cohort 1.) | 3
Cohort 2 (The milestone represents the number of participants in Cohort 2.) | 13
Completed | 15
Not Completed | 1
Not completed — Withdrawal of consent (not due to adverse event) | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug during the treatment period were included in the baseline analysis.
Groups:
- VX-147: All participants received VX-147 at a dosage of 15 mg qd for 2 weeks and VX-147 at a dosage of 45 mg qd for 11 weeks. Part A was enrolled in 2 cohorts: Cohort 1 and Cohort 2. Cohort 1 included participants with urine protein to creatinine ratio (UPCR) approximately ≥3 g/g (± 10%) and <10 g/g and estimated glomerular filtration rate (eGFR) approximately ≥30 mL/min/1.73 m2 (± 10%). Cohort 2 included participants with UPCR approximately ≥0.8 g/g (± 10%) and <2.7 g/g and eGFR approximately ≥30 mL/min/1.73 m2.
Arm/Group | VX-147
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The Baseline data were planned to be presented separately for Cohort 1 and Cohort 2. Here, "Number Analyzed" signifies participants who were evaluable for specified Cohort of the study.
  years
    Cohort 1: number analyzed (Participants) | 3
    Cohort 1 | 45.0 (10.5)
    Cohort 2: number analyzed (Participants) | 13
    Cohort 2 | 37.3 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented separately for Cohort 1 and Cohort 2. Here, "Number Analyzed" signifies participants who were evaluable for specified Cohort of the study.
  Participants
    Cohort 1: number analyzed (Participants) | 3
    Cohort 1: Female | 2
    Cohort 1: Male | 1
    Cohort 2: number analyzed (Participants) | 13
    Cohort 2: Female | 7
    Cohort 2: Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented separately for Cohort 1 and Cohort 2. Here, "Number Analyzed" signifies participants who were evaluable for specified Cohort of the study.
  Participants
    Cohort 1: number analyzed (Participants) | 3
    Cohort 1: Hispanic or Latino | 0
    Cohort 1: Not Hispanic or Latino | 3
    Cohort 1: Unknown or Not Reported | 0
    Cohort 2: number analyzed (Participants) | 13
    Cohort 2: Hispanic or Latino | 0
    Cohort 2: Not Hispanic or Latino | 13
    Cohort 2: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented separately for Cohort 1 and Cohort 2. Here, "Number Analyzed" signifies participants who were evaluable for specified Cohort of the study.
  Participants
    Cohort 1: number analyzed (Participants) | 3
    Cohort 1: American Indian or Alaska Native | 0
    Cohort 1: Asian | 0
    Cohort 1: Native Hawaiian or Other Pacific Islander | 0
    Cohort 1: Black or African American | 3
    Cohort 1: White | 0
    Cohort 1: More than one race | 0
    Cohort 1: Unknown or Not Reported | 0
    Cohort 2: number analyzed (Participants) | 13
    Cohort 2: American Indian or Alaska Native | 0
    Cohort 2: Asian | 0
    Cohort 2: Native Hawaiian or Other Pacific Islander | 0
    Cohort 2: Black or African American | 13
    Cohort 2: White | 0
    Cohort 2: More than one race | 0
    Cohort 2: Unknown or Not Reported | 0
Urine Protein to Creatinine Ratio (UPCR) [Mean (Standard Deviation); unit: g/g] — Population: The baseline data were planned to be presented for the overall treatment arm (i.e. Cohort 1 and Cohort 2). Here, "Number Analyzed" signifies participants who were evaluable for specified Cohort of the study.
  g/g
    Cohort 1: number analyzed (Participants) | 3
    Cohort 1 | 3.47 (1.07)
    Cohort 2: number analyzed (Participants) | 13
    Cohort 2 | 1.77 (0.49)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in UPCR
Time Frame: From Baseline up to Week 13
Population: The Full Analysis Set (FAS) included all participants who received at least 1 dose of study drug in the treatment period. Here "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome and the "Number Analyzed" signifies participants who were evaluable for the specified Cohorts.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Groups:
- VX-147: All participants received VX-147 at a dosage of 15 mg qd for 2 weeks and VX-147 at a dosage of 45 mg qd for 11 weeks and had ≥ 80% adherence to investigational product. Part A was enrolled in 2 cohorts: Cohort 1 and Cohort 2. Cohort 1 included participants with urine protein to creatinine ratio (UPCR) approximately ≥3 g/g (± 10%) and <10 g/g and estimated glomerular filtration rate (eGFR) approximately ≥30 mL/min/1.73 m2 (± 10%). Cohort 2 included participants with UPCR approximately ≥0.8 g/g (± 10%) and <2.7 g/g and eGFR approximately ≥30 mL/min/1.73 m2.
Arm/Group | VX-147
Number analyzed (Participants) | 13
percent change
  Cohort 1: number analyzed (Participants) | 3
  Cohort 1 | -47.7 [-70.1 to -8.5]
  Cohort 2: number analyzed (Participants) | 10
  Cohort 2 | -47.5 [-63.4 to -24.6]
  Total | -47.6 [-60.0 to -31.3]

2. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From Baseline up to Week 17
Population: Safety set included all participants who received at least 1 dose of study drug in the treatment period. Here, the "Number Analyzed" signifies participants who were evaluable for the specified cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | VX-147
Number analyzed (Participants) | 16
Participants
  Cohort 1: Participants With TEAEs: number analyzed (Participants) | 3
  Cohort 1: Participants With TEAEs | 3
  Cohort 1: Participants With SAEs: number analyzed (Participants) | 3
  Cohort 1: Participants With SAEs | 0
  Cohort 2: Participants With TEAEs: number analyzed (Participants) | 13
  Cohort 2: Participants With TEAEs | 12
  Cohort 2: Participants With SAEs: number analyzed (Participants) | 13
  Cohort 2: Participants With SAEs | 1

3. Secondary Outcome: Maximum Observed Concentration (Cmax) of VX-147
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, and 12 hours post-dose on Day 1 and Week 5
Population: The PK set included all those who received at least 1 dose of study drug. Though participants in this study were divided into two cohorts based on their UPCR range, PK data was collected and presented based on dose levels as all participants received 15 mg qd for 2 weeks and 45 mg qd for 11 weeks. Therefore, presenting data based on cohorts as per UPCR range was not relevant for purpose of PK endpoints. Here "Number Analyzed" signifies participants who were evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/ml)
Arm/Group | VX-147
Number analyzed (Participants) | 16
micrograms per milliliter (mcg/ml)
  15 mg qd: Day 1: number analyzed (Participants) | 15
  15 mg qd: Day 1 | 0.168 (0.0630)
  45 mg qd: Week 5: number analyzed (Participants) | 14
  45 mg qd: Week 5 | 0.846 (0.303)

4. Secondary Outcome: Observed Pre-dose Concentration (Ctrough) of VX-147
Time Frame: Pre-dose on Day 8, 15, Week 3, 5, 9 and 13
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | VX-147
Number analyzed (Participants) | 16
mcg/ml
  15 mg qd: Day 8 | 0.153 (0.0984)
  15 mg qd: Day 15: number analyzed (Participants) | 15
  15 mg qd: Day 15 | 0.123 (0.0796)
  45 mg qd: Week 3: number analyzed (Participants) | 15
  45 mg qd: Week 3 | 0.379 (0.249)
  45 mg qd: Week 5: number analyzed (Participants) | 15
  45 mg qd: Week 5 | 0.492 (0.265)
  45 mg qd: Week 9: number analyzed (Participants) | 14
  45 mg qd: Week 9 | 0.446 (0.342)
  45 mg qd: Week 13: number analyzed (Participants) | 13
  45 mg qd: Week 13 | 0.529 (0.302)

5. Secondary Outcome: Area Under the Concentration Time-curve From 0 to 24 Hours (AUC0-24hr) of VX-147
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 12 and 24 hours Post-dose on Week 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour*mcg/mL (h*mcg/mL)
Arm/Group | VX-147
Number analyzed (Participants) | 13
hour*mcg/mL (h*mcg/mL) | 15.3 (6.37)

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 17
Groups:
- VX-147 : Cohort 1: Cohort 1 included participants with urine protein to creatinine ratio (UPCR) approximately ≥3 g/g (± 10%) and <10 g/g and estimated glomerular filtration rate (eGFR) approximately ≥30 mL/min/1.73 m2 (± 10%).
- VX-147: Cohort 2: Cohort 2 included participants with UPCR approximately ≥0.8 g/g (± 10%) and <2.7 g/g and eGFR approximately ≥30 mL/min/1.73 m2
- VX-147 Total: All participants received VX-147 at a dosage of 15 mg qd for 2 weeks and VX-147 at a dosage of 45 mg qd for 11 weeks. Part A was enrolled in 2 cohorts: Cohort 1 and Cohort 2. Cohort 1 included participants with urine protein to creatinine ratio (UPCR) approximately ≥3 g/g (± 10%) and <10 g/g and estimated glomerular filtration rate (eGFR) approximately ≥30 mL/min/1.73 m2 (± 10%). Cohort 2 included participants with UPCR approximately ≥0.8 g/g (± 10%) and <2.7 g/g and eGFR approximately ≥30 mL/min/1.73 m2.
Arm/Group | VX-147 : Cohort 1 | VX-147: Cohort 2 | VX-147 Total
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/13 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/13 | 1/16
Other Adverse Events (participants affected / at risk) | 3/3 | 12/13 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VX-147 : Cohort 1 (N=3) | VX-147: Cohort 2 (N=13) | VX-147 Total (N=16)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VX-147 : Cohort 1 (N=3) | VX-147: Cohort 2 (N=13) | VX-147 Total (N=16)
Palpitations (Cardiac disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 3
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 2
Peripheral swelling (General disorders) | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 1
Tinea pedis (Infections and infestations) | 1 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Blood bicarbonate decreased (Investigations) | 0 | 2 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1
Electrocardiogram ST segment depression (Investigations) | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1
Transaminases increased (Investigations) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 2
Headache (Nervous system disorders) | 1 | 3 | 4
Depressed mood (Psychiatric disorders) | 0 | 1 | 1
Thinking abnormal (Psychiatric disorders) | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT04340362/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT04340362/SAP_001.pdf